CLINICAL TRIAL: NCT00257959
Title: Optimal Pharmacological Therapy In Implantable Defibrillator Patients (OPTIC)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Connolly, Stuart, M.D. (Individual)
Collaborators: Abbott Medical Devices (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1
Record Dates: First submitted 2005-11-22; First posted 2005-11-24 (Estimated); Last update posted 2006-07-27 (Estimated); Status verified 2005-11

CONDITIONS: Ventricular Tachycardia
MeSH Terms: conditions — Tachycardia, Ventricular

INTERVENTIONS:
Drug: amiodarone beta blocker sotalol

SUMMARY:
This is an open parallel design randomized trial of amiodarone plus a beta blocker vs a beta blocker alone vs sotalol for the prevention of ICD shocks in patients receiving an ICD for spontaneous or inducible ventricular tachycardia or fibrillation

ELIGIBILITY:
Inclusion Criteria: spontaneous or inducible ventricular tachycardia or fibrillation -

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400
Dates: Start 2001-01; Study Completion 2004-10

PRIMARY OUTCOMES:
ICD shock for any cause

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Connolly, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

REFERENCES:
- [Result] Connolly SJ, Dorian P, Roberts RS, Gent M, Bailin S, Fain ES, Thorpe K, Champagne J, Talajic M, Coutu B, Gronefeld GC, Hohnloser SH; Optimal Pharmacological Therapy in Cardioverter Defibrillator Patients (OPTIC) Investigators. Comparison of beta-blockers, amiodarone plus beta-blockers, or sotalol for prevention of shocks from implantable cardioverter defibrillators: the OPTIC Study: a randomized trial. JAMA. 2006 Jan 11;295(2):165-71. doi: 10.1001/jama.295.2.165. PMID 16403928
- [Result] Hohnloser SH, Dorian P, Roberts R, Gent M, Israel CW, Fain E, Champagne J, Connolly SJ. Effect of amiodarone and sotalol on ventricular defibrillation threshold: the optimal pharmacological therapy in cardioverter defibrillator patients (OPTIC) trial. Circulation. 2006 Jul 11;114(2):104-9. doi: 10.1161/CIRCULATIONAHA.106.618421. Epub 2006 Jul 3. PMID 16818810